CLINICAL TRIAL: NCT01928927
Title: Effects of Telmisartan on Fibrotic and Inflammatory Contributors to End-Organ Disease in HIV-Infected Patients Well Controlled on Antiretroviral Therapy
Brief Title: Telmisartan to Reduce AIDS-Related Fibrotic and Inflammatory Contributors (TRAFIC Study)
Acronym: TRAFIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5317; UM1AI068636 (NIH)
Record Dates: First submitted 2013-08-22; First posted 2013-08-27 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2020-06

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Telmisartan (Experimental)
  Interventions: Drug: Telmisartan
- Arm B: No Study Drug (No Intervention): Participants received no study drug and followed the week 0-48 evaluation schedule.

INTERVENTIONS:
Drug: Telmisartan — Participants received Telmisartan 40 mg daily during weeks 0-4 followed by telmisartan 80 mg daily during weeks 5-48.
  Arms: Arm A: Telmisartan

SUMMARY:
The main goal of this study was to see if a drug called telmisartan would decrease fibrosis (scarring) and inflammation (irritation) in people who are infected with HIV and doing well on their HIV medications. The study was also done to see what effects telmisartan has on other signs of disease and inflammation in the body, and to see whether people who have HIV can take telmisartan safely and without side effects that make them want to stop the drug. Telmisartan is FDA-approved for treating high blood pressure and decreasing the chance of heart attacks and strokes in people over the age of 55 years of age who are at high risk for these events.

DETAILED DESCRIPTION:
This was a multicenter, randomized, open label, phase IIb, two-arm study to evaluate the effects of telmisartan on fibrotic and inflammatory contributors to end-organ disease in HIV-infected subjects well controlled on antiretroviral therapy (ART). Participants were randomized 2:1 to the telmisartan and control arms. The participants on telmisartan took 40 mg telmisartan daily during weeks 0-4 followed by telmisartan 80 mg daily during weeks 5-48. The participants in the control arm did not take any study medication, but did undergo all evaluations. All participants were followed for 48 weeks after randomization.

The study clinic visits included Step 1 entry, Step 2 entry, and weeks 4, 12, 24, 36, 48. Biopsies for the primary outcomes were collected at Step 1 entry and Week 48. The evaluations of safety (clinical assessment for signs and symptoms, diagnoses, laboratory tests) were done at Step 2 entry and weeks 4, 12, 24, 36, 48.

The co-primary objectives assessed the effects of telmisartan for 48weeks on lymph node and adipose tissue collagen I deposition.

Currently, the results are entered for the primary outcome measures only. The results on the secondary outcomes will be posted when they become available.

ELIGIBILITY:
Step 1 Inclusion Criteria:

* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to Step 1 entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, or plasma HIV-1 RNA viral load >2000 copies/mL on two occasions.
* On antiretroviral therapy (ART) continuously for ≥48 weeks prior to Step 1 entry.
* Documentation of HIV-1 RNA <50 copies/mL at screening, performed by any US laboratory that has a CLIA certification or its equivalent.
* At least one HIV-1 RNA level <200 copies/mL in the 48 weeks prior to Step 1 entry (not including the screening).
* No change in ART regimen in the 12 weeks prior to Step 1 entry (except as noted below).

NOTE: Modifications of ART dosing during the 12 weeks prior to Step 1 entry are permitted. In addition, the change in formulation (eg, from standard formulation to fixed dose combination or single tablet regimen) is allowed within 12 weeks of Step 1 entry. A within-class single drug substitution (eg, switch from nevirapine to efavirenz or from atazanavir to darunavir) is allowed within 12 weeks of Step 1 entry, with the exception of a switch from any other NRTI to abacavir. No other changes in ART in the 12 weeks prior to Step 1 entry are permitted.

* No active plan to change ART for the 48-week study duration.
* Body mass index (BMI) 20-35 kg/m^2.
* For females of reproductive potential, negative serum or urine pregnancy test within 3 days prior to Step 1 entry.
* Ability and willingness of subject or legal guardian/representative to provide informed consent.
* Willingness to undergo the Step 1 entry and week 48 lymphoid and adipose tissue biopsies.

Step 2 Inclusion Criteria:

* Entry lymphoid tissue and adipose tissue specimen for assay of the primary endpoint has been obtained. (Prior to Letter of Amendment #2, 11/19/14)
* (Letter of Amendment #2, 11/19/14) Entry lymphoid tissue and adipose tissue specimens for assay of the primary endpoint have been obtained, entered into the ACTG's Laboratory Data Management System (LDMS), and confirmed by the protocol team as adequate for endpoint determination.

NOTE: If the lymph node specimen is determined by the protocol team to be inadequate for endpoint determination despite the interventions summarized in LOA #2, the participant will be permitted to enroll if adequate adipose tissue is obtained. However, as change in lymph node fibrosis remains one of the primary endpoints of this study, it is critical that every effort be made to obtain an adequate sample while still trying to minimize complication rates.

* Willingness to undergo the week 48 lymphoid and adipose tissue biopsies. (Prior to Letter of Amendment #2, 11/19/14)
* (Letter of Amendment #2, 11/19/14) Willingness to undergo the week 48 lymphoid and adipose tissue biopsies.

NOTE: A week 48 lymph node biopsy is not required if the Step 1 lymph node specimen was deemed inadequate as noted in 4.3.1. Week 48 adipose tissue biopsies will still be required for these participants.

Step 1 Exclusion Criteria:

* More than one HIV-1 RNA >200 copies/mL in the 48 weeks prior to Step 1 entry.
* One HIV-1 RNA 200-500 copies/mL in the 24 weeks prior to Step 1 entry that is not immediately preceded and followed by HIV-1 RNA <50 copies/mL.

NOTE: The preceding viral load <50 copies/mL may be >24 weeks prior to Step 1 entry.

* Confirmed systolic blood pressure >160 mmHg or <100 mmHg or diastolic blood pressure >100 mmHg.
* Known untreated renal artery stenosis.
* Known cirrhosis or severe liver disease (eg, ascites, encephalopathy, history of variceal bleeding).

NOTE: Potential subjects with chronic hepatitis B or C virus infection with no known cirrhosis or severe liver disease may participate in the study, provided there are no plans to start therapy for hepatitis C infection during the 48-week study duration.

* Unstable coronary artery disease/angina or decompensated congestive heart failure.
* Either breastfeeding or pregnant within 24 weeks prior to Step 1 entry.
* Use of thiazolidinediones or any angiotensin receptor blocker (ARB) or angiotensin converting enzyme inhibitor (ACEi) in the 24 weeks prior to Step 1 entry. If the subject took either of these classes of medications for less than 2 weeks in the 24 weeks prior to Step 1 entry, the subject may enroll if 30 days have passed since the last dose. If the subject is diabetic and/or has a calculated glomerular filtration rate (GFR) <60mL/min, aliskiren-containing medications are also prohibited.
* History of intolerance, other than cough, to any ARB or ACEi.
* Use of anticoagulants other than aspirin 81 mg or 325 mg daily. NOTE: If the subject is on aspirin 81 mg or 325 mg daily and is willing/able to stop therapy for 7 days prior to the biopsy procedures, the subject may enroll.
* Any known bleeding disorder or coagulopathy.
* Projected need for daily potassium supplementation for ≥2 weeks during the study period.
* The following laboratory values obtained within 30 days prior to Step 1 entry by any US laboratory that has a CLIA certification or its equivalent:

  * Absolute neutrophil count (ANC) ≤750 cells/mm^3
  * Hemoglobin ≤10 g/dL
  * Platelet count ≤75,000/mm^3
  * Calculated creatinine clearance (CrCl) <50 mL/min, as estimated by the Cockcroft-Gault equation
  * Aspartate aminotransferase (AST) (SGOT) >/=3x ULN (upper limit of normal)
  * Alanine aminotransferase (ALT) (SGPT) >/=3x ULN
  * Partial thromboplastin time (PTT) >1.2x ULN
  * Prothrombin time (PT) >1.2x ULN
* Heritable connective tissue disorders (eg Ehlers-Danlos syndrome, osteogenesis imperfecta, Stickler syndrome, Marfan's syndrome).

NOTE: Subjects with acquired/autoimmune chronic inflammatory diseases/connective tissue disorders who are clinically stable (in the opinion of the site investigator) and not on a prohibited medication may enroll with approval of the A5317 study chairs.

* Serious illness requiring systemic treatment and/or hospitalization until subject either completes therapy or is clinically stable on therapy, in the opinion of the site investigator, for at least 7 days prior to Step 1 entry.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Any condition that, in the opinion of the site investigator, would compromise the subject's ability to participate in the study.

Step 2 Exclusion Criteria:

- Any AE associated with the Step 1 entry biopsy that would exclude the subject from undergoing follow-up biopsy at week 48.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan E. Lake, MD, MSc, Study Chair — The University of Texas Health Science Center, Houston; Netanya Sandler, MD, Study Chair — The University of Texas Medical Branch, Galveston
Locations (12):
- United States (11):
  - UCLA CARE Center CRS (601), Los Angeles, California
  - University of Colorado Hospital CRS (6101), Aurora, Colorado
  - Massachusetts General Hospital ACTG CRS (101), Boston, Massachusetts
  - Washington U CRS (2101), St Louis, Missouri
  - University of Rochester Adult HIV Therapeutic Strategies Network CRS (31787), Rochester, New York
  - Unc Aids Crs (3201), Chapel Hill, North Carolina
  - Univ. of Cincinnati CRS (2401), Cincinnati, Ohio
  - Case CRS (2501), Cleveland, Ohio
  - Vanderbilt Therapeutics CRS (3652), Nashville, Tennessee
  - Houston AIDS Research Team CRS (31473), Houston, Texas
  - University of Washington AIDS CRS (1401), Seattle, Washington
- Puerto Rico-AIDS CRS (5401), San Juan, Puerto Rico

REFERENCES:
- See also: The DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009) — http://rsc.tech-res.com/clinical-research-sites/safety-reporting/daids-grading-tables
- Available data/document: Grading table — https://rsc.tech-res.com/clinical-research-sites/safety-reporting/daids-grading-tables

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 58 participants enrolled to Step 1 between January 6, 2014 and April 13, 2015. Step 1 was a run-in period to ensure successful pre-randomization biopsies were obtained. 44 participants did have successful Step 1 biopsy and were randomized to Step 2 between January 13, 2014 and April 22, 2015.
Pre-assignment Details: All participants enrolled to Step 1. Participants with successful Step 1 biopsies and eligible for Step 2 were randomized to the two study arms using a 2:1 allocation ratio with permuted blocks of size 3 and without institutional balancing. There was no stratification.
Groups:
- Arm A: Telmisartan: Participants will receive Telmisartan 40 mg daily during weeks 0-4 followed by telmisartan 80 mg daily during weeks 5-48.
  Telmisartan
- Arm B: No Study Drug: Participants will receive no study drug and will follow week 0-48 evaluation schedule.
  Control
Period: Overall Study
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Started | 29 | 15
Completed | 27 | 14
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: All Step 2 randomized participants with data available for specific measures.
Groups:
- Arm A: Telmisartan: Participants received Telmisartan 40 mg daily during weeks 0-4 followed by telmisartan 80 mg daily during weeks 5-48.
  Telmisartan
- Arm B: No Study Drug: Participants received no study drug and were followed week 0-48 evaluation schedule.
  Control
- Total: Total of all reporting groups
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug | Total
Number analyzed (Participants) | 29 | 15 | 44
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 [41 to 51] | 50 [39 to 52] | 48 [41 to 52]
Age, Customized [Count of Participants; unit: Participants]
  18-29 years | 0 | 2 | 2
  30-39 years | 6 | 2 | 8
  40-49 years | 12 | 3 | 15
  50-59 years | 11 | 6 | 17
  60-69 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 27 | 14 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 1 | 8
  Not Hispanic or Latino | 22 | 14 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 22 | 7 | 29
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 16 | 6 | 22
  Black Non-Hispanic | 5 | 8 | 13
  Hispanic (Regardless of Race) | 7 | 1 | 8
  More than one race | 1 | 0 | 1
IV drug history [Count of Participants; unit: Participants]
  No History | 25 | 13 | 38
  Previous History | 4 | 2 | 6
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 25.4 [23.3 to 29.8] | 23.7 [21.4 to 26.6] | 25.0 [22.6 to 28.4]
Waist circumference [Median (Inter-Quartile Range); unit: cm] — Population: Participants with non-missing waist circumference data.
  cm
    number analyzed (Participants) | 28 | 14 | 42
    (all) | 92 [85 to 100] | 86 [81 to 96] | 88 [84 to 99]
Waist-to-hip ratio [Median (Inter-Quartile Range); unit: ratio] — Population: Participants with non-missing waist circumference data.
  ratio
    number analyzed (Participants) | 28 | 14 | 42
    (all) | 0.94 [0.91 to 0.98] | 0.91 [0.86 to 0.95] | 0.93 [0.89 to 0.97]
CD4+ [Median (Inter-Quartile Range); unit: cells/mm^3] — Population: Participants with non-missing CD4+ data.
  cells/mm^3
    number analyzed (Participants) | 28 | 15 | 43
    (all) | 604 [438 to 812] | 556 [444 to 906] | 588 [444 to 841]
HIV-1 RNA [Count of Participants; unit: Participants]
  <40 copies/ml | 24 | 11 | 35
  40 - <200 copies/ml | 3 | 3 | 6
  >= 200 copies/ml | 2 | 1 | 3
Lymphoid Tissue Collagen I Deposition [Median (Inter-Quartile Range); unit: percent area stain positive] — Population: Participants with non-missing lymphoid tissue collagen I deposition data.
  percent area stain positive
    number analyzed (Participants) | 24 | 15 | 39
    (all) | 15.3 [6.5 to 22.1] | 12.6 [10.3 to 19.1] | 13.9 [8.4 to 20.8]
Adipose Tissue Collagen I Deposition [Median (Inter-Quartile Range); unit: percent area stain positive] | 1.51 [0.54 to 2.69] | 2.83 [1.36 to 4.53] | 2.11 [0.63 to 3.45]

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent Collagen I Deposition on Lymph Node Pathology From Baseline to Week 48
Description: Percent collagen I deposition is defined as the average % collagen stained in multiple uniform sized high magnification images in each sample. Change was absolute change defined as the Week 48 value minus the baseline value.
Time Frame: baseline and week 48
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing lymphoid tissue collagen I deposition.
Measure: Median (Inter-Quartile Range); unit: percent area stain positive
Groups:
- Arm B: No Study Drug: Participants received no study drug and will follow week 0-48 evaluation schedule.
  Control
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 17 | 12
percent area stain positive | -2.44 [-10.60 to 3.77] | -6.08 [-11.66 to 5.84]
Statistical Analysis 1: Comparison: Arm A: Telmisartan vs Arm B: No Study Drug; Null hypothesis: theta = 0.50; Test type: Superiority; p = 0.97, Theta statistic; DeLong & Clarke-Pearson — No adjustment for multiple comparisons; Theta statistic = 0.50, 95% CI 2-sided [0.26 to 0.73] — The theta statistic estimates the probability that a randomly selected outcome from the telmisartan arm is <= a randomly selected outcome from the control arm

2. Primary Outcome: Change in Percent Collagen I Deposition on Subcutaneous Abdominal Adipose Tissue Pathology From Baseline to Week 48
Description: Percent collagen I deposition defined as percentage of fibrotic/collagen area to total area. Change was absolute change defined as the Week 48 value minus the baseline value.
Time Frame: baseline and week 48
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing subcutaneous abdominal adipose tissue collagen I deposition.
Measure: Median (Inter-Quartile Range); unit: percent area stain positive
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 16 | 9
percent area stain positive | -1.43 [-10.61 to 4.17] | 0.36 [-6.57 to 6.41]
Statistical Analysis 1: Comparison: Arm A: Telmisartan vs Arm B: No Study Drug; Null hypothesis: theta = 0.50; Test type: Superiority; p = 0.61, Theta statistic; DeLong & Clarke-Pearson — No adjustment for multiple comparisons; Theta statistic = 0.57, 95% CI 2-sided [0.31 to 0.83] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change in Percent Fibronectin Deposition on Lymph Node Pathology From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing lymphoid tissue fibronectin deposition.
Measure: Median (Inter-Quartile Range); unit: percent area stain positive
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 19 | 11
percent area stain positive | 0.01 [-0.40 to 0.35] | 0.61 [-0.09 to 1.40]

4. Secondary Outcome: Change in Percent Fibronectin Deposition on Subcutaneous Abdominal Adipose Tissue Pathology From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing adipose tissue fibronectin deposition.
Measure: Median (Inter-Quartile Range); unit: percent area stain positive
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 22 | 12
percent area stain positive | -0.82 [-4.00 to 0.45] | -4.01 [-6.02 to -1.63]

5. Secondary Outcome: Change in Percent Collagen VI Deposition on Subcutaneous Abdominal Adipose Tissue Pathology From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing adipose collagen VI deposition.
Measure: Median (Inter-Quartile Range); unit: percent area stain positive
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 22 | 12
percent area stain positive | -0.41 [-4.03 to 0.31] | -1.36 [-2.04 to -0.67]

6. Secondary Outcome: Highest Grade Non-biopsy-related Adverse Event
Description: Safety was summarized as the highest grade non-biopsy-related sign/symptom, laboratory event, or diagnosis per participant.
  Grading (Grade 0: normal, Grade 1: mild, Grade 2: moderate, Grade 3: severe, Grade 4: life-threatening) was done by site clinicians using DAIDS AE Grading table.
  NOTE: As adipose tissue and lymph node biopsies are generally considered to be minimal risk procedures, biopsy safety profile were not formally be evaluated as an endpoint in this protocol.
Time Frame: after baseline to week 48
Population: All Step 2 participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 29 | 15
Participants
  Grade 0 | 12 | 6
  Grade 1 | 0 | 0
  Grade 2 | 11 | 3
  Grade 3 | 5 | 5
  Grade 4 | 1 | 1

7. Secondary Outcome: Change in IL-6 From Baseline to Week 4
Description: Absolute change was calculated as the value at week 4 minus the value at baseline.
Time Frame: baseline and week 4
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing IL-6.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 12
pg/ml | -0.50 [-0.80 to 0.11] | -0.01 [-0.29 to 0.27]

8. Secondary Outcome: Change in IL-6 From Baseline to Week 24
Description: Absolute change was calculated as the value at week 24 minus the value at baseline.
Time Frame: baseline and week 24
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 12
pg/ml | -0.53 [-0.69 to 0.04] | 0.04 [-0.48 to 0.85]

9. Secondary Outcome: Change in IL-6 From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 22 | 13
pg/ml | -0.46 [-0.86 to 0.13] | -0.03 [-0.48 to 1.18]

10. Secondary Outcome: Change in IL-7 From Baseline to Week 4
Description: Absolute change was calculated as the value at week 4 minus the value at baseline.
Time Frame: baseline and week 4
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing IL-7.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 12
pg/ml | 0.48 [-0.21 to 2.18] | -0.32 [-4.34 to 0.37]

11. Secondary Outcome: Change in IL-7 From Baseline to Week 24
Description: Absolute change was calculated as the value at week 24 minus the value at baseline.
Time Frame: baseline and week 24
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 12
pg/ml | 0.51 [-0.13 to 2.32] | -1.36 [-3.94 to 0.44]

12. Secondary Outcome: Change in IL-7 From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 22 | 13
pg/ml | 0.06 [-0.82 to 1.73] | 0.53 [-1.18 to 2.28]

13. Secondary Outcome: Change in Adiponectin From Baseline to Week 4
Description: Absolute change was calculated as the value at week 4 minus the value at baseline.
Time Frame: baseline and week 4
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing adiponectin.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 12
ng/ml | 177.20 [-1624.50 to 1949.70] | 161.00 [-528.30 to 1597.35]

14. Secondary Outcome: Change in Adiponectin From Baseline to Week 24
Description: Absolute change was calculated as the value at week 24 minus the value at baseline.
Time Frame: baseline and week 24
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 12
ng/ml | -582 [-1709.30 to 714.20] | 1222.60 [-867.60 to 3278.15]

15. Secondary Outcome: Change in Adiponectin From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 22 | 13
ng/ml | -138.70 [-1935.20 to 1521.70] | 113.80 [-3150.00 to 907.80]

16. Secondary Outcome: Change in Collagen I C-terminal Pro-peptide (CICP) From Baseline to Week 4
Description: Absolute change was calculated as the value at week 4 minus the value at baseline.
Time Frame: baseline and week 4
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing CICP.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 13
ng/ml | -2.14 [-14.94 to 8.45] | -9.10 [-27.38 to 14.29]

17. Secondary Outcome: Change in Collagen I C-terminal Pro-peptide (CICP) From Baseline to Week 24
Description: Absolute change was calculated as the value at week 24 minus the value at baseline.
Time Frame: baseline and week 24
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 12
ng/ml | -13.78 [-37.69 to 5.93] | -1.17 [-24.43 to 40.16]

18. Secondary Outcome: Change in Collagen I C-terminal Pro-peptide (CICP) From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: as for outcome 16
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 22 | 13
ng/ml | -10.76 [-40.50 to 27.78] | -6.10 [-31.99 to 6.36]

19. Secondary Outcome: Change in Hyaluronic Acid From Baseline to Week 4
Description: Absolute change was calculated as the value at week 4 minus the value at baseline.
Time Frame: baseline and week 4
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing hyaluronic acid.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 12
ng/ml | -0.03 [-8.46 to 16.63] | 3.14 [-7.29 to 14.42]

20. Secondary Outcome: Change in Hyaluronic Acid From Baseline to Week 24
Description: Absolute change was calculated as the value at week 24 minus the value at baseline.
Time Frame: baseline and week 24
Population: as for outcome 19
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 12
ng/ml | -1.62 [-18.32 to 1.19] | 3.71 [-5.83 to 30.20]

21. Secondary Outcome: Change in Hyaluronic Acid From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: as for outcome 19
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 22 | 13
ng/ml | -2.74 [-18.52 to 9.84] | -1.79 [-6.96 to 14.49]

22. Secondary Outcome: Change in sCD14 From Baseline to Week 4
Description: Absolute change was calculated as the value at week 4 minus the value at baseline.
Time Frame: baseline and week 4
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing sCD14.
Measure: Median (Inter-Quartile Range); unit: mcg/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 12
mcg/ml | -0.03 [-0.37 to 0.08] | 0.05 [-0.06 to 0.25]

23. Secondary Outcome: Change in sCD14 From Baseline to Week 24
Description: Absolute change was calculated as the value at week 24 minus the value at baseline.
Time Frame: baseline and week 24
Population: as for outcome 22
Measure: Median (Inter-Quartile Range); unit: mcg/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 12
mcg/ml | 0.06 [-0.19 to 0.26] | -0.08 [-0.15 to 0.09]

24. Secondary Outcome: Change in sCD14 From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: as for outcome 22
Measure: Median (Inter-Quartile Range); unit: mcg/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 22 | 13
mcg/ml | -0.08 [-0.26 to 0.12] | 0 [-0.17 to 0.36]

25. Secondary Outcome: Change in sCD163 From Baseline to Week 4
Description: Absolute change was calculated as the value at week 4 minus the value at baseline.
Time Frame: baseline and week 4
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing sCD163.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 12
ng/ml | 34.08 [-33.96 to 174.04] | 0.88 [-45.16 to 106.08]

26. Secondary Outcome: Change in sCD163 From Baseline to Week 24
Description: Absolute change was calculated as the value at week 24 minus the value at baseline.
Time Frame: baseline and week 24
Population: as for outcome 25
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 12
ng/ml | 58.72 [-44.52 to 206.52] | 9.58 [-49.40 to 56.72]

27. Secondary Outcome: Change in sCD163 From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: as for outcome 25
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 22 | 13
ng/ml | 31.14 [-200.04 to 160.20] | 5.32 [-117.80 to 96.84]

28. Secondary Outcome: Change in TGF-β1 From Baseline to Week 4
Description: Absolute change was calculated as the value at week 4 minus the value at baseline.
Time Frame: baseline and week 4
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing TGF-β1.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 12
pg/ml | 793.37 [-2080.11 to 3877.98] | -1074.87 [-5328.36 to 603.32]

29. Secondary Outcome: Change in TGF-β1 From Baseline to Week 24
Description: Absolute change was calculated as the value at week 24 minus the value at baseline.
Time Frame: baseline and week 24
Population: as for outcome 28
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 12
pg/ml | 175.02 [-1249.67 to 4478.09] | 678.43 [-3983.91 to 2816.12]

30. Secondary Outcome: Change in TGF-β1 From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: as for outcome 28
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 22 | 13
pg/ml | -319.17 [-3429.94 to 1203.98] | -516.45 [-2307.66 to 2090.85]

31. Secondary Outcome: Change in TGF-β2 From Baseline to Week 4
Description: Absolute change was calculated as the value at week 4 minus the value at baseline.
Time Frame: baseline and week 4
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing TGF-β2.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 12
pg/ml | 70.74 [-135.73 to 147.97] | -129.40 [-272.80 to -5.13]

32. Secondary Outcome: Change in TGF-β2 From Baseline to Week 24
Description: Absolute change was calculated as the value at week 24 minus the value at baseline.
Time Frame: baseline and week 24
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 12
pg/ml | 75.84 [-39.61 to 134.71] | -134.68 [-345.89 to -8.64]

33. Secondary Outcome: Change in TGF-β2 From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 22 | 13
pg/ml | 44.45 [-201.77 to 164.44] | -55.94 [-201.52 to 119.60]

34. Secondary Outcome: Change in TGF-β3 From Baseline to Week 4
Description: Absolute change was calculated as the value at week 4 minus the value at baseline.
Time Frame: baseline and week 4
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing TGF-β3.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 12
pg/ml | 31.26 [-39.82 to 254.89] | -95.17 [-450.42 to -10.83]

35. Secondary Outcome: Change in TGF-β3 From Baseline to Week 24
Description: Absolute change was calculated as the value at week 24 minus the value at baseline.
Time Frame: baseline and week 24
Population: as for outcome 34
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 12
pg/ml | 34.64 [-16.14 to 226.95] | -68.01 [-341.55 to 101.57]

36. Secondary Outcome: Change in TGF-β3 From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: as for outcome 34
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 22 | 13
pg/ml | -0.47 [-176.53 to 175.68] | -55.21 [-163.05 to 135.04]

37. Secondary Outcome: Change in Circulating CD4+ T Cell Count From Baseline to Week 12
Description: Absolute change was calculated as the value at week 12 minus the value at baseline.
Time Frame: baseline and week 12
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing CD4+ count.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 20 | 10
cells/mm^3 | -17.50 [-133 to 26] | 59.50 [-24 to 108]

38. Secondary Outcome: Change in Circulating CD4+ T Cell Count From Baseline to Week 24
Description: Absolute change was calculated as the value at week 24 minus the value at baseline.
Time Frame: baseline and week 24
Population: as for outcome 37
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 20 | 12
cells/mm^3 | 13 [-55 to 95] | 61.5 [-16.5 to 186.5]

39. Secondary Outcome: Change in Circulating CD4+ T Cell Count From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: as for outcome 37
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 13
cells/mm^3 | 9 [-24 to 45] | 97 [4 to 111]

40. Secondary Outcome: Change in Circulating CD8+ T Cell Count From Baseline to Week 12
Description: Absolute change was calculated as the value at week 12 minus the value at baseline.
Time Frame: baseline and week 12
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing CD8+ count.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 20 | 10
cells/mm^3 | -33.5 [-130 to 111.5] | 83 [30 to 154]

41. Secondary Outcome: Change in Circulating CD8+ T Cell Count From Baseline to Week 24
Description: Absolute change was calculated as the value at week 24 minus the value at baseline.
Time Frame: baseline and week 24
Population: as for outcome 40
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 20 | 12
cells/mm^3 | -3.5 [-97 to 103.5] | 80.5 [-8 to 181.5]

42. Secondary Outcome: Change in Circulating CD8+ T Cell Count From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: as for outcome 40
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 13
cells/mm^3 | 10 [-72 to 101] | 97 [-24 to 169]

43. Secondary Outcome: Change in Fasting Glucose From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing fasting glucose.
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 13
mg/dl | 4 [-3 to 8] | 2 [-5 to 12]

44. Secondary Outcome: Change in Fasting HDL Cholesterol From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing fasting HDL cholesterol.
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 13
mg/dl | -1 [-6 to 1] | -4 [-7 to 6]

45. Secondary Outcome: Change in Fasting Insulin From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing fasting insulin.
Measure: Median (Inter-Quartile Range); unit: uIU/ml
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 22 | 13
uIU/ml | 3 [-1 to 4] | 0 [-2 to 8]

46. Secondary Outcome: Change in Fasting LDL Cholesterol From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing fasting LDL cholesterol.
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 13
mg/dl | -12 [-30.2 to 12] | -7.4 [-20.6 to 18.8]

47. Secondary Outcome: Change in Fasting Total Cholesterol From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing fasting total cholesterol.
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 13
mg/dl | -8 [-23 to 4] | -2 [-8 to 9]

48. Secondary Outcome: Change in Fasting Triglycerides From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing fasting triglycerides.
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 13
mg/dl | 7 [-23 to 29] | -16 [-23 to 63]

49. Secondary Outcome: Change in HOMA-IR From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing HOMA-IR.
Measure: Median (Inter-Quartile Range); unit: (mg/dl)x(uIU/ml)/405
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 13
(mg/dl)x(uIU/ml)/405 | 0.76 [-0.02 to 1.01] | -0.04 [-0.42 to 1.03]

50. Secondary Outcome: Prevalence of Metabolic Syndrome at Week 24.
Description: Components of the metabolic syndrome will be defined according to the 2004 updated National Cholesterol Education Program Adult Treatment Panel III [NCEP ATP III] criteria) as the presence of any 3 of the following: Waist: >40" (101.6 cm) in men, >35" (88.9 cm) in women with the exception of Asian-Americans: >35" (88.9 cm) in men, 31" (78.7 cm) in women; Fasting HDL-C <40 mg/dL in men, <50 mg/dL in women; Fasting TG ≥150 mg/dL; Diastolic blood pressure ≥85 mmHg or systolic blood pressure ≥130 mmHg; Fasting plasma glucose ≥100 mg/dL.
  NOTE: This definition of metabolic syndrome may be subject to change in accordance with current guidelines at the time of the final analysis. It will be defined in the Final Statistical Analysis Plan prior to data review for final analysis.
Time Frame: Week 24
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing metabolic syndrome components.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 11
Participants
  Metabolic syndrome | 6 | 1
  No metabolic syndrome | 15 | 10

51. Secondary Outcome: Presence of Metabolic Syndrome at Week 48.
Description: Components of the metabolic syndrome were defined according to the 2004 updated National Cholesterol Education Program Adult Treatment Panel III [NCEP ATP III] criteria) as the presence of any 3 of the following: Waist: >40" (101.6 cm) in men, >35" (88.9 cm) in women with the exception of Asian-Americans: >35" (88.9 cm) in men, 31" (78.7 cm) in women; Fasting HDL-C <40 mg/dL in men, <50 mg/dL in women; Fasting TG ≥150 mg/dL; Diastolic blood pressure ≥85 mmHg or systolic blood pressure ≥130 mmHg; Fasting plasma glucose ≥100 mg/dL.
Time Frame: Week 48
Population: as for outcome 50
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 13
Participants
  Metabolic syndrome | 7 | 0
  No metabolic syndrome | 14 | 13

52. Secondary Outcome: Change in Waist Circumference From Baseline to Week 24
Description: Absolute change was calculated as the value at week 24 minus the value at baseline.
Time Frame: baseline and week 24
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing waist circumference.
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 20 | 10
cm | 0.90 [-0.15 to 3.40] | 0.57 [-3.87 to 5.80]

53. Secondary Outcome: Change in Waist Circumference From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: as for outcome 52
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 12
cm | 0.77 [-2.03 to 2.93] | -0.08 [-4.95 to 5.05]

54. Secondary Outcome: Change in Waist-to-hip Ratio From Baseline to Week 24
Description: Absolute change was calculated as the value at week 24 minus the value at baseline.
Time Frame: baseline and week 24
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing waist-to-hip ratio.
Measure: Median (Inter-Quartile Range); unit: waist cm : hip cm
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 20 | 10
waist cm : hip cm | 0 [-0.01 to 0.03] | 0.01 [0 to 0.03]

55. Secondary Outcome: Change in Waist-to-hip Ratio From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: baseline and week 48
Population: as for outcome 54
Measure: Median (Inter-Quartile Range); unit: waist cm : hip cm
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 21 | 11
waist cm : hip cm | 0 [-0.01 to 0.02] | 0.02 [-0.02 to 0.04]

56. Secondary Outcome: Change in Expression of CD38+HLA-DR+ on CD4+ From Baseline to Week 24
Description: Absolute change was calculated as the value at week 24 minus the value at baseline.
Time Frame: 24 weeks
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing CD4+CD38+HLA-DR+ data.
Measure: Median (Inter-Quartile Range); unit: Percent of CD4+ expressing CD38+HLA-DR+
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 19 | 12
Percent of CD4+ expressing CD38+HLA-DR+ | 0.20 [-0.60 to 1.50] | -1.35 [-2.10 to -0.75]

57. Secondary Outcome: Change in Expression of CD38+HLA-DR+ on CD8+ From Baseline to Week 24
Description: Absolute change was calculated as the value at week 24 minus the value at baseline.
Time Frame: 24 weeks
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing CD8+CD38+HLA-DR+ data.
Measure: Median (Inter-Quartile Range); unit: Percent of CD8+ expressing CD38+HLA-DR+
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 19 | 12
Percent of CD8+ expressing CD38+HLA-DR+ | 0.60 [-0.60 to 3.00] | -0.95 [-2.10 to -0.40]

58. Secondary Outcome: Change in Expression of CD38+HLA-DR+ on CD4+ From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: 48 weeks
Population: as for outcome 56
Measure: Median (Inter-Quartile Range); unit: Percent of CD4+ expressing CD38+HLA-DR+
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 20 | 13
Percent of CD4+ expressing CD38+HLA-DR+ | -0.30 [-0.90 to 1.10] | -0.60 [-1.30 to 0.20]

59. Secondary Outcome: Change in Expression of CD38+HLA-DR+ on CD8+ From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: 48 weeks
Population: as for outcome 57
Measure: Median (Inter-Quartile Range); unit: Percent of CD8+ expressing CD38+HLA-DR+
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 20 | 13
Percent of CD8+ expressing CD38+HLA-DR+ | -0.40 [-1.55 to 0.85] | -0.20 [-1.80 to 0.90]

60. Secondary Outcome: Change in Expression of CD163+ in Adipose Tissue From Baseline to Week 48
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: 48 weeks
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing CD163+ adipose tissue data.
Measure: Median (Inter-Quartile Range); unit: Percent of CD163+ adipose tissue cells
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 20 | 12
Percent of CD163+ adipose tissue cells | -0.19 [-5.55 to 3.76] | 0.87 [-2.52 to 2.75]

61. Secondary Outcome: Change in Expression of CD4+ in Lymphoid Tissue From Baseline to Week 48.
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: 48 weeks
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing CD4+ lymphoid tissue data.
Measure: Median (Inter-Quartile Range); unit: Percent of CD4+ lymphoid tissue cells
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 11 | 6
Percent of CD4+ lymphoid tissue cells | 1 [-5.2 to 3.7] | -7.8 [-12.3 to 2.1]

62. Secondary Outcome: Change in Expression of CD8+ in Lymphoid Tissue From Baseline to Week 48.
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: 48 weeks
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing CD8+ lymphoid tissue data.
Measure: Median (Inter-Quartile Range); unit: Percent of CD8+ lymphoid tissue cells
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 11 | 6
Percent of CD8+ lymphoid tissue cells | -1.19 [-5.3 to 1.5] | 3.9 [1.0 to 9.2]

63. Secondary Outcome: Change in Expression of CD163+ in Lymphoid Tissue From Baseline to Week 48.
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: 48 weeks
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing CD163+ lymphoid tissue data.
Measure: Median (Inter-Quartile Range); unit: Percent of CD163+ lymphoid tissue cells
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 11 | 6
Percent of CD163+ lymphoid tissue cells | -0.13 [-0.81 to 0.81] | 0.15 [-0.77 to 0.69]

64. Secondary Outcome: Change in Expression of CD68+ in Lymphoid Tissue From Baseline to Week 48.
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: 48 weeks
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing CD68+ lymphoid tissue data.
Measure: Median (Inter-Quartile Range); unit: Percent of CD68+ lymphoid tissue cells
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 11 | 6
Percent of CD68+ lymphoid tissue cells | -0.02 [-0.48 to 0.49] | 0.08 [-1.07 to 0.24]

65. Secondary Outcome: Change in Expression of CD38+HLA-DR+ on CD4+ in Lymphoid Tissue From Baseline to Week 48.
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: 48 weeks
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing CD38+HLA-DR+ on CD4+ lymphoid tissue data.
Measure: Median (Inter-Quartile Range); unit: Percent of CD38+HLA-DR+ on CD4+ cells
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 11 | 6
Percent of CD38+HLA-DR+ on CD4+ cells | -0.33 [-2.55 to 0.87] | 0.06 [-0.35 to 1.11]

66. Secondary Outcome: Change in Expression of CD38+HLA-DR+ on CD8+ in Lymphoid Tissue From Baseline to Week 48.
Description: Absolute change was calculated as the value at week 48 minus the value at baseline.
Time Frame: 48 weeks
Population: Per-protocol population: Participants who 1) completed the protocol, 2) completed treatment (if on telmisartan arm), 3) did not have confirmed virologic failure, 4) had paired biopsies at baseline and week 48.
  Additionally, have non-missing CD38+HLA-DR+ on CD8+ lymphoid tissue data.
Measure: Median (Inter-Quartile Range); unit: Percent of CD38+HLA-DR+ on CD8+ cells
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
Number analyzed (Participants) | 11 | 6
Percent of CD38+HLA-DR+ on CD8+ cells | 0.13 [-3.95 to 0.63] | -0.22 [-0.72 to 0.48]

ADVERSE EVENTS:
Time Frame: From baseline to Week 48.
Description: Protocol definition of Other (Not Including Serious) Adverse Events: 1) signs and symptoms Grade ≥2 and any that led to a change in treatment regardless of grade; 2) all new diagnoses; 3) Grade ≥2 lab values. All lab toxicities that led to a change in treatment or were associated with a diagnosis were recorded, regardless of grade. The following labs regardless of grade: creatinine, AST, ALT, hemoglobin, platelet count, fasting lipids and fasting glucose. DAIDS AE Grading Table (V1.0) was used.
Arm/Group | Arm A: Telmisartan | Arm B: No Study Drug
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/15
Serious Adverse Events (participants affected / at risk) | 3/29 | 1/15
Other Adverse Events (participants affected / at risk) | 24/29 | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Telmisartan (N=29) | Arm B: No Study Drug (N=15)
Angina unstable (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Herpes zoster disseminated (Infections and infestations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Telmisartan (N=29) | Arm B: No Study Drug (N=15)
Eye pruritus (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1
Anorectal swelling (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 0
Perianal erythema (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1
Rectal discharge (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 2 | 0
Peripheral swelling (General disorders) | 2 | 0
Pyrexia (General disorders) | 3 | 0
Seasonal allergy (Immune system disorders) | 0 | 1
Gastroenteritis shigella (Infections and infestations) | 2 | 0
Perirectal abscess (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 4 | 1
Aspartate aminotransferase increased (Investigations) | 4 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 4 | 2
Blood cholesterol increased (Investigations) | 13 | 4
Blood creatinine increased (Investigations) | 2 | 1
Blood glucose increased (Investigations) | 4 | 1
Blood magnesium decreased (Investigations) | 2 | 1
Blood phosphorus decreased (Investigations) | 7 | 3
Blood sodium decreased (Investigations) | 7 | 2
Low density lipoprotein increased (Investigations) | 13 | 4
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 2 | 0
Weight decreased (Investigations) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Sleep disorder (Psychiatric disorders) | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Penile discharge (Reproductive system and breast disorders) | 0 | 1
Penile pain (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No